CLINICAL TRIAL: NCT02751801
Title: Health Burden of Hypophosphatasia
Status: Completed | Type: Observational
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: STH19182
Record Dates: First submitted 2016-04-01; First posted 2016-04-26 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Hypophosphatasia
MeSH Terms: conditions — Hypophosphatasia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adults and children with hypophosphatasia: Healthcare use interview
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention

SUMMARY:
Hypophosphatasia (HPP) is a genetic disorder caused by mutation in the tissue-non-specific alkaline phosphatase gene (TNSALP). It causes impaired bone mineralisation, fractures, tooth loss, muscle weakness and possibly other adverse health outcomes.

The infantile-onset forms are severe, and were often fatal until the recent availability of a treatment (Asfotase Alfa). The childhood-onset forms are less severe, and the adult-onset form is mild, and often unrecognised or misdiagnosed as osteoporosis.

The less severe forms of the disease are not well described, and because there has been no available treatment there has not been much research in adults. However, now that treatment is available there is a possibility of a clinical trial in adults. To know whether there is a need for a trial there is a need to determine if there is a significant personal and economic burden associated with the less severe forms of HPP.

The study consists of a clinical interview and notes review of adults and children with confirmed (by biochemical and genetic testing) HPP attending metabolic bone clinics in Sheffield to establish their clinical problems and healthcare use. There are currently about 26 adults and 8 children attending clinics in Sheffield.

The information will be used to plan a data search and health economic analysis of the burden of HPP from the UK Clinical Practice Research Database in collaboration with Pharmatelligence (a healthcare data group based within the University of Cardiff).

DETAILED DESCRIPTION:
This is an observational retrospective study to describe the clinical problems and healthcare use of adults and children with hypophosphatasia.

Interviews will be conducted with patients with childhood- and adult-onset hypophosphatasia (and the parents of the children). Hospital notes, appointment records and GP summary care records will also be reviewed.

These sources will be used to describe their clinical problems, how these problems affect their daily function, and which healthcare services they have used.

Patients will attend for a single visit to obtain informed consent and conduct the interview.

Health problems specifically assessed in detail will include:

* Fractures
* Dental problems
* Skeletal complications
* Mobility problems
* Neurosurgical complications
* Seizures
* Respiratory complications
* Depression and anxiety
* Side effects of treatment including hypercalcaemia and hyperphosphataemia Deaths will also be recorded

Health care resource assessment will include

* Primary care episodes
* Secondary and tertiary care outpatient episodes
* In-patient episodes
* Nutritional support
* Therapy support
* Dental treatment
* Over the counter medication use

A case data report form will be developed as an iterative process through the period of the interviews to ensure that all data of potential interest is captured. Because the condition is not well described it is important that the data reported is not limited to the areas where it might be already expected to find problems.

ELIGIBILITY:
Inclusion Criteria:

* Hypophosphatasia

Exclusion Criteria:

* Unable/unwilling to give informed consent

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults and children with hypophosphatasia
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2016-11; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
description of healthcare use | one day study visit
  Descriptive data on which health care services the patient has used in relation to HPP

SECONDARY OUTCOMES:
healthcare use appointments | one day study visit
  descriptive data on number of healthcare encounters
healthcare cost | one day study visit
  estimated healthcare cost attributable to HPP

CONTACTS AND LOCATIONS:
Overall Officials: Richard Eastell, MD FRCP, Principal Investigator — University of Sheffield
Locations (1):
- Academic Unit of Bone Metabolism (Sheffield), Sheffield, South Yorks, United Kingdom